CLINICAL TRIAL: NCT00391183
Title: Effect of Palliative Biliary Stenting Versus Conservative Treatment on the Quality of Life (QOL) of Patients With Unresectable Carcinoma of the Gallbladder With Hiliar Block: A Randomised Controlled Trial
Brief Title: Palliative Biliary Stenting on the Quality of Life of Patients With Unresectable Carcinoma Gallbladder With Hiliar Block.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Pramod Kumar Garg, Additional Professor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GE-CAGB/2005
Record Dates: First submitted 2006-10-19; First posted 2006-10-23 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Gallbladder Cancer
Keywords: Gallbladder cancer; Quality of life; Stenting; Survival; Performance status
MeSH Terms: conditions — Gallbladder Neoplasms

ARMS (2):
- Endoscopic stenting (Active Comparator): patients with biliary obstruction will undergo endoscopic stenting.
  Interventions: Procedure: Biliary stenting
- Best supportive care (No Intervention)

INTERVENTIONS:
Procedure: Biliary stenting — ERCP and stenting
  Arms: Endoscopic stenting

SUMMARY:
The purpose of the study is to determine whether palliative biliary stenting improves the quality of life, of gallblader cancer patients, who present with hilar block and obstructive jaundice.

DETAILED DESCRIPTION:
For most patients with gallbladder cancer, cure is not possible and treatment should be therefore aimed at palliation of symptoms and maintaining quality of life (QOL) in the few months between diagnosis and death. Most of these patients suffer from intractable pruritis, pain, anorexia and general debility. Biliary stenting leads to a reduction in pruritis and jaundice, and is commonly offered to many unresectable patients. However stenting related complications like cholangitis, rescue percutaneous treatment and need for prolonged hospitalization often impair the remaining short survival of these patients. In these patients improving the QOL should be the primary focus, and survival a secondary end point in disease management. No study has addressed the issue of QOL of patients with gallbladder cancer, post stenting.

Three clinical studies have evaluated the change in the QOL of patients with malignant biliary obstruction after of endoscopic stenting. Ballinger et al evaluated 19 patients with unresectable pancreatic carcinoma before stenting and upto 12 weeks or death after stenting. The Rotterdam Symptom Checklist and the Hospital Anxiety and Depression Scale were used. Significant improvements were seen in the parameters of mood, indigestion, appetite and level of activity. Luman et al studied 47 inoperable patients with malignant biliary strictures. The European Organisation for Research and Treatment of Cancer QOL questionnaire (EORTC QLQ-C30) was used at baseline and 1 month after stenting. For patients successfully completing the follow up, significant improvement in emotional, cognitive , and global health scores was found after stenting. In addition to the expected improvement in pruritis and jaundice , anorexia, diarrhea and sleep pattern were also improved. Abraham et al studied 50 patients with malignant biliary obstruction without liver metastasis considered non surgical candidates, and undergoing palliative biliary stenting. The SF-36 Health Survey Questionnaire was used to quantify QOL at baseline and 1 month after stent insertion. Follow up data was available for only 26 patients. Among these patients a significant reduction in the bilirubin level was associated with improvement in the social function and mental health. A high baseline bilirubin (> 14mg/dL) was associated with a lack of improvement at 1 month follow up.

Hence existing data regarding improvement in the QOL of patients undergoing palliative biliary stenting is sparce and incomplete. Gallbladder cancer presenting a hilar block is the most common biliary malignancy in India. Hilar tumors are associated with more technical failure of stenting, higher cholangitis rates, earlier stent blockage, and shorter survival as compared to distal biliary tumors. Only 6 patients with Klatskin tumors were included in one of the study.8 Patients with hilar block were either not included6, or were not specified7 in the other studies.

Health related quality of life (QOL) refers to the impact of a medical condition or its treatment on a person's expected physical, psychological and social well being.

Calman states that QOL evaluations measure the difference between the "hopes and expectations" of an individual and that individual's present experience.

The multidimensionality that is commonly assessed in QOL measures includes

1. Physical symptoms of the disease or its treatment or concurrent illness.
2. Functional capacity (ability and energy) for daily routine, social interactions, intellectual activity, emotional reactions and adjustments, economic independence.
3. Self-perception of wellness or its absence. There are two basic types of instruments for measuring the QOL: generic and disease specific. Generic instruments focus on the main components that constitute QOL, and are intended to be applied in a wide range of populations and health states across all diseases. There are many excellent validated self-completion questionnaires for cancer patients eg. EORTC QOL questionnaire, Functional assessment of Cancer Therapy (FACT), Rotterdam Symptom Checklist (RSCL), Functional Living Index Cancer (FLIC). All these questionnaires are multidimensional, and it is rarely required to develop a new instrument.

The EORTC QLQ-C30 has been developed in a multi-cultural setting, and translations are available in 43 languages. The instrument has been shown to be valid, reliable, and responsive to change. Disease specific modules are available to supplement the core questionnaire. Reference data is available for calculating sample size. The questionnaire is easily understood by most patients and is quick to complete (mean time 11 minutes).

The EORTC QLQ-C30 is a 30- item questionnaire composed of multi-item scales and single items that reflects the multidimensionality of the quality of life construct. It incorporates five functional scales (physical, role, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), and a global health and quality of life scale. The remaining single items assess additional symptoms commonly reported by cancer patients (dyspnea, appetite loss, sleep disturbance, constipation and diarrhea), as well as the perceived financial impact of the disease and its treatment. The functional scales have 16 questions, symptom scales have 6 questions, global quality of life has two questions, and there are six single item questions. For ease of interpretation, all scale and item scores are linearly transformed to a 0 to 100 scale. For the 5 functional scales and the global quality of life scale, a higher score represents a better level of functioning. For the symptom oriented scales and items, a higher score corresponds to a higher level of symptoms.

Hence we plan to prospectively study unresectable gallbladder cancer patients with hilar block to evaluate whether palliative stenting improves their quality of life, and whether the benefit afforded outweighs the early and late complications of stenting.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with unresectable gallbladder cancer (Bismuth type II to IV).
2. Eastern Cooperative Oncology Group Performance (ECOG) status 0-3.

Exclusion Criteria:

1. Preoperative stenting
2. ECOG status 4
3. Distant residence precluding follow up visits, or unwillingness to return for follow up.
4. Poor comprehension of the Hindi QOL questionnaire.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Improvement in the physical functioning scale (containing five items) of EORTC QLQ-30 one month after after biliary stenting. | 30 days

SECONDARY OUTCOMES:
Improvements in other functional and social scales and single items of EORTC QLQ-30 | 30 days
Survival | 30 days
Hospital stay | 30 days
Cost of therapy | 30 days
Complications | 30 days
Performance status change | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Pramod Garg, M.D, D.M., Study Director — All India Institute of Medical Sciences; Vikram Bhatia, M.D, D.M., Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medical Sciences, New Delhi, India

REFERENCES:
- [Background] Ballinger AB, McHugh M, Catnach SM, Alstead EM, Clark ML. Symptom relief and quality of life after stenting for malignant bile duct obstruction. Gut. 1994 Apr;35(4):467-70. doi: 10.1136/gut.35.4.467. PMID 7513672
- [Background] Luman W, Cull A, Palmer KR. Quality of life in patients stented for malignant biliary obstructions. Eur J Gastroenterol Hepatol. 1997 May;9(5):481-4. doi: 10.1097/00042737-199705000-00013. PMID 9187881
- [Background] Abraham NS, Barkun JS, Barkun AN. Palliation of malignant biliary obstruction: a prospective trial examining impact on quality of life. Gastrointest Endosc. 2002 Dec;56(6):835-41. doi: 10.1067/mge.2002.129868. PMID 12447294